CLINICAL TRIAL: NCT06134830
Title: Clinical Outcome and Quality of Life in Differentiated Thyroid Cancer Patients Treated With Different Doses of Radioactive Iodine.
Brief Title: Differentiated Thyroid Cancer Patients Treated With Different Doses of Radioactive Iodine.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hager Hamdy Sayed Mohammed, Clinical outcome and quality of life in differentiated thyroid cancer patients treated with different doses of radioactive iodine., Assiut University
Other Study IDs: thyroid cancer and RAI
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: RAI — Radioactive iodine

SUMMARY:
1. Determine the frequency of utilizing single and multiple doses of radioactive iodine (RAI) in treatment of differentiated thyroid cancer.
2. Asses the impact of various doses of radioactive iodine on the management of differentiated thyroid cancer.
3. Investigate the influence of thyroid cancer on the quality of life of affected patients.

DETAILED DESCRIPTION:
Differentiated thyroid cancer represents more than 90% of cancer thyroid [1]. Total thyroidectomy is considered the mainstay of curative therapy, with radioactive iodine (RAI) in order to ablate or treat remnant thyroid tissue in the surgical bed and/or elsewhere [2]. The two main objectives for treatment of differentiated cancer thyroid are reducing the probability of cancer recurrence and facilitating serological surveillance via thyroglobulin (TG). The 2015 American Thyroid Association (ATA) guidelines as well as European Consensus Conference described three main risk stratification for thyroid cancer including: low, intermediate and high risk [3] [4]. According to the 2015 ATA guidelines, low- dose (1110 MBq) 131I ablation is recommended for low-to- intermediate-risk patients, while high-dose (3700 MBq or more) 131I ablation may be required for high-risk patients to remove microscopic residual disease(4). The optimal RAI activity needed to achieve the best objective RAI response and to minimize RAI specific adverse effects is not known since there are many factors that should be considered while determining the dose including age of the patient and many pathological factors [5, 6]. Therefore, dose adjustment might be needed for patients with same risk classification. Just following the guidelines might not be optimal for treatment of individual differentiated thyroid cancer [5]. Accordingly, in our centre the administrated activities are varied among our clinicians. In this study, we aim to retrospective analyse patients with differentiated thyroid cancer received variable (single and multiple) doses of RAI in each risk group and to assess their clinical outcome. As thyroid cancer has a very good prognosis, there a debate that quality of life may be affected in patients with high risk compared to low and intermediate risks. Additionally, we intend to evaluate the impact of thyroid cancer on quality of life by questionnaire filled by patients with different risk groups.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with differentiated cancer thyroid either papillary or follicular underwent total thyroidectomy with or without lymph node dissection.

  * Available data of patients' records.

Exclusion Criteria:

* • Missed follow up data.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with differentiated cancer thyroid treated at Assiut University Hospitals.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with differentiated thyroid cancer receiving a single dose of RAI. | 2 Years
  Proportion of differentiated thyroid cancer patients treated with single dose of RAI.

SECONDARY OUTCOMES:
Quality of life score of affected patients will be assessed through validated quality of life questionnaire (SF-36). | 2 Years
  Questionnaire for quality of life in differentiated thyroid cancer patients.

REFERENCES:
- [Background] Pacini F, Fuhrer D, Elisei R, Handkiewicz-Junak D, Leboulleux S, Luster M, Schlumberger M, Smit JW. 2022 ETA Consensus Statement: What are the indications for post-surgical radioiodine therapy in differentiated thyroid cancer? Eur Thyroid J. 2022 Jan 1;11(1):e210046. doi: 10.1530/ETJ-21-0046. PMID 34981741
- [Background] Andresen NS, Buatti JM, Tewfik HH, Pagedar NA, Anderson CM, Watkins JM. Radioiodine Ablation following Thyroidectomy for Differentiated Thyroid Cancer: Literature Review of Utility, Dose, and Toxicity. Eur Thyroid J. 2017 Jul;6(4):187-196. doi: 10.1159/000468927. Epub 2017 Mar 23. PMID 28868259
- [Background] Pacini F, Schlumberger M, Dralle H, Elisei R, Smit JW, Wiersinga W; European Thyroid Cancer Taskforce. European consensus for the management of patients with differentiated thyroid carcinoma of the follicular epithelium. Eur J Endocrinol. 2006 Jun;154(6):787-803. doi: 10.1530/eje.1.02158. No abstract available. PMID 16728537
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967